CLINICAL TRIAL: NCT01451281
Title: Evaluation of Skeletal Muscle, Cardiac, and Diaphragm Imaging Biomarkers for GSK2402968 Effects in Ambulatory Boys With Duchenne Muscular Dystrophy
Brief Title: Studying Skeletal Muscle, Heart, and Diaphragm Imaging in Boys With Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110261; 11-N-0261
Record Dates: First submitted 2011-10-08; First posted 2011-10-13 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05-20

CONDITIONS: Muscular Dystrophy; Muscular Disease
Keywords: Ultrasonography; Muscular Dystrophy; Neuromuscular Disease; Oligonucleotide; Magnetic Resonance Imaging (MRI); Duchenne Muscular Dystrophy; DND
MeSH Terms: conditions — Muscular Dystrophies; Muscular Diseases; Neuromuscular Diseases; Muscular Dystrophy, Duchenne

SUMMARY:
Background:

- Duchenne muscular dystrophy (DMD) is a disease in which the muscles are unable to make the protein dystrophin. Without this protein, the muscles become gradually weaker. A new medicine called GSK2402968 is being tested to see if it can help prevent or slow down this loss of muscle strength. In this study, boys with DMD and healthy volunteers will have different types of imaging studies to see which ones provide the best images of the muscles. This information will help researchers use these imaging techniques to test the safety and effectiveness of GSK2402968 and other agents.

Objectives:

- To test magnetic resonance imaging and ultrasound techniques that can detect changes in muscles of boys with DMD.

Eligibility:

* Boys who have DMD and are in the GSK2402968 drug test study.
* Healthy boys of the same age as the above study participants.

Design:

* Participants will be screened with a medical history and physical exam.
* Healthy volunteers will have one 2-hour visit with three tests. Magnetic resonance imaging (MRI) scans of the skeletal muscles and heart and diaphragm muscles will be carried out. Muscle ultrasound imaging of leg and arm muscles will also be done. Participants should not perform heavy physical activity like school sports or long walks during the week before the visit.
* Participants in the GSK2402968 study will have the same series of tests as the healthy volunteers. The tests will be given during the study screening phase. They will be repeated after 3 months and 6 months of receiving the study agent (GSK2402968 or placebo) and at 6 months after stopping the GSK study.

DETAILED DESCRIPTION:
Objective:

Duchenne muscular dystrophy (DMD) is the most frequent inherited fatal childhood disease. Antisense oligonucleotide (AON)-induced exon skipping is a promising therapeutic strategy for DMD that is currently being explored in clinical trials. Magnetic resonance imaging (MRI) and ultrasound imaging methods are sensitive to key processes in dystrophic muscle such as edema and fat infiltration and therefore could serve as a biomarker of disease progression and therapeutic response. Our objective is to explore the potential of these imaging biomarkers for GSK2402968 (AON) effects in ambulatory boys with DMD. The primary objective is to assess longitudinal changes in skeletal muscle structural MRI measures reflecting fat and edema in the lower extremities in ambulatory boys with DMD receiving GSK2402968 or placebo

Study Population:

We aim to enroll up to 65 ambulatory boys with DMD. Healthy volunteer/control boys (up to 25) matched for the age-range will be recruited to obtain pilot data for imaging studies.

Design:

This prospective study of skeletal muscle, cardiac, and diaphragm imaging at the NIH will be offered to all subjects participating in a phase 2, double blind, exploratory parallel-group, placebo-controlled clinical study in ambulatory subjects with DMD resulting from a mutation that can be corrected by exon 51 skipping induced by GSK2402968 (parent study; DMD114876). Subjects will travel with a family member to the NIH for MRI and ultrasound assessments during the screening phase of the parent study or up to 3 weeks after randomization and additionally at the following time points in the parent study: at 12 weeks ( 3 weeks), and 24 weeks ( 3 weeks) during the blinded treatment period; and finally, after completion of 24 week post-treatment phase (at 48 weeks 4 weeks). If not randomized, the subjects will have a one-time evaluation during the screening phase of the parent study. Pilot data also will be obtained from healthy boys (matched for the age-range) for comparisons to allow exploration of MRI and ultrasound measures specific to pathology in the ambulatory boys with DMD. Subjects will not be treated with GSK2402968 or any other experimental drug at the NIH. There are no follow-up or termination procedures for this study.

Outcome Measures:

Primary Outcome Measure: MRI changes in skeletal muscle percent fat in the lower extremities using T1w GRE Dixon method at 24 weeks from baseline in the parent study in ambulatory boys with DMD receiving GSK2402968 or placebo. Secondary outcome measures: Differences in the following outcome measures between healthy boys and ambulatory boys with DMD at baseline; and changes in these measures over time in the parent study at 12 weeks, 24 weeks, and 48 weeks from baseline in ambulatory boys with DMD receiving GSK2402968 or placebo: 1. Skeletal muscle MRI: relative muscle fat/water quantified by T1w GRE Dixon imaging method in skeletal muscles; Muscle edema assessed by T2 imaging; Muscle fat/water content and edema additionally quantified by IDEAL-CPMG method; and 2. Cardiac MRI: Cardiac function (ejection fraction/ LV function) assessed by SSFP Cine MRI and manual planimetry of LV volumes and mass at end systole and end diastole; Myocardial fat content assessed by Multiecho Dixon Fat /Water Separation method; Myocardial edema assessed by T2 quantification; Myocardial T1 assessed by MOLLI (modified Look-Locker Inversion recovery).

Exploratory Outcome Measures: MRI changes in muscle architecture and water diffusivity will be assessed by Diffusion EPI MRI. If well tolerated, then we will use a portable device (Ankle IntelliStretch device, RehabTek) to study the effects of exercise on selected MRI measures in leg muscles. Muscle ultrasound will be used to monitor changes in skeletal muscle volume, echogenicity and stiffness. Dynamic breathing MRI will be performed to measure diaphragm motion during free breathing and voluntary maximal inspiration and exhalation.

ELIGIBILITY:
* INCLUSION CRITERIA:

DMD Subjects

* Eligible for the parent study
* Willing and able to comply with all protocol requirements and procedures, including MRI without sedation
* Able to give informed assent and parent(s)/legal guardian to give informed consent in writing signed by the subject and/or parent(s)/legal guardian

Healthy Volunteers

* Must be unaffected by a neuromuscular condition
* Willing and able to comply with all protocol requirements and procedures, including MRI without sedation.
* Able to give informed assent and parent(s)/legal guardian to give informed consent in writing signed by the subject and/or parent(s)/legal guardian.

EXCLUSION CRITERIA:

DMD Subjects and Healthy Volunteers

* Having metal objects in his body that are not MRI-safe. These include the following objects: 1) pacemakers or other implanted electrical devices; 2) brain stimulators; 3) some types of dental implants; 4) aneurysm clips (metal clips on the wall of a large artery); 5) metallic prostheses (including metal pins and rods, heart valves, and cochlear implants; 6) implanted delivery pump; 7) permanent eye liner; or 8) shrapnel fragments.
* Having a fear of closed spaces

Ages: 5 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2011-09-15; Study Completion 2019-05-20

PRIMARY OUTCOMES:
Changes in muscle fat content quantified by T1w GRE Dixon imaging method in skeletal muscles in the lower extremities at 24 weeks from baseline in the parent study in ambulatory boys with DMD receiving GSK2402968 or placebo

SECONDARY OUTCOMES:
Changes in muscle edema by T2w imaging and muscle fat/water content by IDEAL-CPMG method; myocardial fat/edema and cardiac function by MRI methods in DMD boys receiving GSK2402968 or placebo as well as DMD boys at baseline versus healthy volunte...
Changes in water diffusivity by MRI; muscle volume, fat, and fibrosis by ultrasound; and diaphragm function by dynamic breathing MRI methods in DMD boys receiving GSK2402968 or placebo as well as DMD boys at baseline versus healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Fischbeck, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aartsma-Rus A, Van Deutekom JC, Fokkema IF, Van Ommen GJ, Den Dunnen JT. Entries in the Leiden Duchenne muscular dystrophy mutation database: an overview of mutation types and paradoxical cases that confirm the reading-frame rule. Muscle Nerve. 2006 Aug;34(2):135-44. doi: 10.1002/mus.20586. PMID 16770791
- [Background] Goemans NM, Tulinius M, van den Akker JT, Burm BE, Ekhart PF, Heuvelmans N, Holling T, Janson AA, Platenburg GJ, Sipkens JA, Sitsen JM, Aartsma-Rus A, van Ommen GJ, Buyse G, Darin N, Verschuuren JJ, Campion GV, de Kimpe SJ, van Deutekom JC. Systemic administration of PRO051 in Duchenne's muscular dystrophy. N Engl J Med. 2011 Apr 21;364(16):1513-22. doi: 10.1056/NEJMoa1011367. Epub 2011 Mar 23. PMID 21428760
- [Background] Hoffman EP, Brown RH Jr, Kunkel LM. Dystrophin: the protein product of the Duchenne muscular dystrophy locus. Cell. 1987 Dec 24;51(6):919-28. doi: 10.1016/0092-8674(87)90579-4. PMID 3319190